CLINICAL TRIAL: NCT00279942
Title: Effect of Revival Soy on Fibromyalgia Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Physicians Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2155-05
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Dietary Supplements; Rheumatologic Diseases; Complementary and Alternative Medicine
MeSH Terms: conditions — Fibromyalgia | interventions — Isoflavones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy (Active Comparator): A shake that contained 20 g of soy protein and 160 mg of soy isoflavone.
  Interventions: Dietary Supplement: Soy
- Placebo (Placebo Comparator): A shake that contained 20 g of milk-based protein (casein) and no isoflavone.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Soy — Drink a shake (vanilla and chocolate taste) once a day for 6 weeks.
  Other Names: Isoflavone
  Arms: Soy
Other: Placebo — Drink a shake (vanilla and chocolate taste) once a day for 6 weeks.
  Arms: Placebo

SUMMARY:
Fibromyalgia is characterized by widespread pain that can lead to significant patient dysfunction and economic burden to society. The management of patients with fibromyalgia is difficult and no single treatment modality has been successful. We propose to study the effect of dietary soy supplement on quality of life associated with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia syndrome is a chronic, generalized pain syndrome that affects the musculoskeletal system (1). This syndrome is typically diagnosed in patients who experience generalized musculoskeletal pain and have excessive tenderness in at least 11 of 18 specific points (2). Although the primary cause of fibromyalgia syndrome is unclear, a growing body of evidence indicates that the widespread pain associated with this syndrome is due to abnormalities in the central nervous system. Therefore, drug therapy for fibromyalgia syndrome is most often aimed at the central nervous system and includes tricyclic antidepressants, selective serotonin reuptake inhibitors, dual serotonin and norepinephrine reuptake inhibitors, analgesics, and anticonvulsants (1).

In addition to medical therapies, complementary and alternative medicine therapies have been used to treat fibromyalgia syndrome symptoms (3). Soy is a widely used dietary supplement that has not been previously tested for treating fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Women and men age 18 - 76
* Able to understand and sign a consent form
* Able to participate fully in all aspects of the study
* Currently participating in Mayo Clinic's Fibromyalgia Treatment Program

Exclusion Criteria:

* Pregnant or lactating women
* Allergy to soy or other study product ingredients
* Diagnosis of bipolar disorder, schizophrenia or dementia
* Diagnosis of diabetes mellitus or inflammatory bowel disease
* Presently on soy product or use of soy within the last 30 days

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To gather preliminary data on whether dietary soy supplement can improve quality of life in patients with fibromyalgia as measured by the Fibromyalgia Impact Questionnaire (FIQ) and the Center for Epidemiologic Studies Depression Scale (CES-D). | 6 Weeks

SECONDARY OUTCOMES:
To assess the feasibility of recruiting 50 patients with fibromyalgia into a study of using a dietary supplement. | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Goldenberg DL, Burckhardt C, Crofford L. Management of fibromyalgia syndrome. JAMA. 2004 Nov 17;292(19):2388-95. doi: 10.1001/jama.292.19.2388. PMID 15547167
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Holdcraft LC, Assefi N, Buchwald D. Complementary and alternative medicine in fibromyalgia and related syndromes. Best Pract Res Clin Rheumatol. 2003 Aug;17(4):667-83. doi: 10.1016/s1521-6942(03)00037-8. PMID 12849718
- [Result] Wahner-Roedler DL, Thompson JM, Luedtke CA, King SM, Cha SS, Elkin PL, Bruce BK, Townsend CO, Bergeson JR, Eickhoff AL, Loehrer LL, Sood A, Bauer BA. Dietary soy supplement on fibromyalgia symptoms: a randomized, double-blind, placebo-controlled, early phase trial. Evid Based Complement Alternat Med. 2011;2011:350697. doi: 10.1093/ecam/nen069. Epub 2011 Jun 23. PMID 18990724
- See also: Revival Soy — http://www.revivalsoy.com/